CLINICAL TRIAL: NCT00883545
Title: The Effect of a Woman Endoscopist on Adherence to Screening Colonoscopy in Women
Brief Title: Study of Adherence to Colonoscopy in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 08-1045; NCT00903097 (obsolete NCT alias)
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2012-09

CONDITIONS: Colonoscopy
Keywords: Adherence to screening colonoscopy in women

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Woman endoscopist (Experimental)
  Interventions: Other: Woman endoscopist
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Woman endoscopist — This group will receive an invitation to schedule a screening colonoscopy with a woman endoscopist.
  Arms: Woman endoscopist
Other: Usual care — This group will receive an invitation to schedule a screening colonoscopy with any available endoscopist.
  Arms: Usual care

SUMMARY:
The purpose of this study is to determine whether women who are offered screening colonoscopy will be more likely to schedule and complete this procedure if they are given the option of a woman endoscopist.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third leading cause of cancer death in women. Although there are a variety of options for colon cancer screening, colonoscopy is thought to be the best modality for women. Despite recommendations by multiple societies, adherence to CRC screening among women is suboptimal. One possible barrier to adherence may be the gender of the endoscopist. Recent studies have shown that a large proportion of surveyed women would prefer a woman endoscopist. These studies suggest that having the option of a woman endoscopist would increase adherence to colonoscopy; however, there is no published literature that addresses this question.

Hypothesis

Women who are offered screening colonoscopy will be more likely to schedule and complete this procedure if they are given the option of a woman endoscopist.

Specific Aims

Primary

* Determine whether the option of a woman endoscopist is associated with increased woman patient adherence to screening colonoscopy.
* Assess the proportion of women who request a woman endoscopist when this option is made available to them.

Secondary

* Identify socio-demographic predictors of (a) completing a screening colonoscopy and (b) requesting a woman endoscopist (e.g. race/ethnicity, age, health insurance, marital status).

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age between 50 and 70
* Receiving primary care at a University Medicine clinic

Exclusion Criteria:

* No visit to a University Medicine clinic in 18 months or more
* Deceased
* Pregnant
* Terminal or cancer diagnosis
* No longer receiving primary care at a University Medicine clinic

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Determine whether the option of a woman endoscopist is associated with increased woman patient willingness to schedule and complete screening colonoscopy. | 6 months

SECONDARY OUTCOMES:
Identify socio-demographic predictors of (a) completing a screening colonoscopy and (b) requesting a woman endoscopist (e.g. race/ethnicity, age, health insurance, marital status). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Denberg, MD, PhD, Principal Investigator — University of Colorado Denver Health Sciences Center
Locations (1):
- University of Colorado Denver Health Sciences Center, Aurora, Colorado, United States